CLINICAL TRIAL: NCT05605808
Title: Impact of Aerobic Training Combed With Diet Protocol on Immune System in Post Mastectomy Patients Receiving Chemotherapy
Brief Title: Aerobic Training and Diet on the Immune System in Postmastectomy Patients Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003747
Record Dates: First submitted 2022-10-08; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Immune Deficiency; Diet, Healthy; Breast Cancer
Keywords: Aerobic exercises; Diet therapy; Immune function; Mastectomy
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The model is composed of the aerobic and diet protocol group (Group A), the diet protocol group (Group B), and the aerobic training group (Group C).
Who Masked: Outcomes Assessor
Masking Description: Computer randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercises and diet protocol group (Experimental): The participant will be managed by aerobic exercise by using a treadmill, two times per week. Its intensity was equivalent to 60-85% of each patient's maximum heart rate and lasted 20 minutes in the first week and 30 minutes after the second week in addition to the diet protocol specific diet designed to boost the immune system through edible seeds and nuts which are rich in proteins, fats, fibers, minerals, and vitamins for twelve weeks.
  Interventions: Other: Aerobic exercises; Other: Diet protocol
- Diet protocol group (Active Comparator): The participant will be managed by a specific diet protocol designed to boost the immune system through edible seeds and nuts which are rich in proteins, fats, fibers, minerals, and vitamins for twelve weeks.
  Interventions: Other: Diet protocol
- Aerobic exercises group (Active Comparator): The participant will be managed by aerobic exercise by using a treadmill, two times per week. Its intensity was equivalent to 60-85% of each patient's maximum heart rate and lasted 20 minutes in the first week and 30 minutes after the second week for twelve weeks as a total treatment time.
  Interventions: Other: Aerobic exercises

INTERVENTIONS:
Other: Aerobic exercises — Aerobic exercise by using the treadmill, two times per week. Its intensity was equivalent to 60-85% of each patient's maximum heart rate and lasted 20 minutes in the first week and 30 minutes in weeks 2-12.
  Arms: Aerobic exercises and diet protocol group; Aerobic exercises group
Other: Diet protocol — A specific diet for three months is designed to boost the immune system through edible seeds and nuts which are rich in proteins, fats, fibers, minerals, and vitamins.
  Arms: Aerobic exercises and diet protocol group; Diet protocol group

SUMMARY:
The purpose of the study was to investigate the impact of aerobic exercise combined with diet protocol on the immune system in post-mastectomy patients receiving chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy reduces circulating lymphocytes levels, which affect lymphocytes in breast cancer patients during the therapy itself or up to 3 months after the last chemotherapy cycle, so the study is developed to investigate the impact of aerobic exercise combined with diet protocol on the immune system in post-mastectomy patients receiving chemotherapy. Sixty post-mastectomy women were receiving chemotherapy and aged from 40-60 years selected from the outpatient clinic of the oncology department in the New Cairo hospital in the Police Academy. They will be assigned randomly into three equal groups, the aerobic exercises and diet protocol group, the diet protocol group, and the aerobic exercises group. The immunological markers; total lymphocyte count (TLC), neutrophil-to-lymphocyte ratio(NLR), and platelet-to-lymphocyte ratio(PLR) will be measured at baseline and after twelve weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female post-mastectomy patients.
* Age range is between 40-60 years old.
* All patients will enter the study after having their informed consent.
* All patients are undergoing chemotherapy treatment with AC protocol (Adriamycin with endoxan) for four cycles (every 21 days ).
* All patients have finished the first stage of chemotherapy treatment

Exclusion Criteria:

* Cardiac disease patients.
* Uncontrolled hypertension patients.
* Patients with thyroid disease.
* Patients with lymphatic complications.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients
Enrollment: 60 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-02-21 (Estimated); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
The change in total lymphocyte count. | Baseline and twelve weeks after the intervention.
  from patient's blood sample analysis for immunological markers in lab.
The change in neutrophil to lymphocyte ratio. | Baseline and twelve weeks after the intervention.
  from patient's blood sample analysis for immunological markers in lab.
The change in platelet to lymphocyte ratio. | Baseline and twelve weeks after the intervention.
  from patient's blood sample analysis for immunological markers in lab.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA Elsayeh, PhD, Study Director — Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No